CLINICAL TRIAL: NCT00088283
Title: A Phase II Randomized, Dose-Ranging, Double-Masked, Multi-Center Trial, in Parallel Groups, Determining Safety, Efficacy and PK of Intravitreous Injections of Pegaptanib Sodium Compared to Sham Injection for 30 Weeks in Patients With Recent Vision Loss Due to Macular Edema Secondary to CRVO
Brief Title: Pegaptanib Sodium Compared to Sham Injection in Patients With Recent Vision Loss Due to Macular Edema Secondary to Central Retinal Vein Occlusion (CRVO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP 1011B
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: Retinal Vein Occlusion
Keywords: CRVO; Central Retinal Vein Occlusion; RVO; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium

SUMMARY:
Eyetech Pharmaceuticals Inc. and Pfizer, Inc. are studying an investigational drug, MacugenTM, for the possible treatment of CRVO. An investigational drug is one that has not been approved by the U.S. Food and Drug Administration (FDA). This investigational drug may slow the growth of abnormal blood vessels in the eye and may reduce tissue swelling in the eye.

The purpose of this study is to compare the safety and efficacy of a Macugen™ injection to a "pretend" injection. In addition, the purpose of this study is to measure the action of the study drug in the body over a period of time and to check for the presence of the study drug in your blood (called pharmacokinetics or PK).

This study will involve approximately 90 people. People who decide to participate will have an equal chance (1 in 3) to receive one of three study injections, two of which are Macugen™ and one of which is a "pretend" injection.

DETAILED DESCRIPTION:
This study will consist of 3 phases: a screening phase which will last up to two weeks, a confirmation phase which will last one day, and a randomization phase (the patient will be assigned by chance to a study group in this phase) which will last approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* CRVO must have occurred within the past 6 months and be associated with macular edema determined by OCT.
* Vision in the study eye corresponding to between approximately 20/50 to 20/400 and better than or equal to approximately 20/200 in the fellow eye.

Exclusion Criteria:

* Presence of signs of old branch retinal vein occlusion (BRVO) or CRVO in the study eye or any other retinal vascular disease including diabetic retinopathy.
* Vitreous hemorrhage except breakthrough hemorrhage from intraretinal hemorrhage.
* Prior pan retinal photocoagulation (PRP) or sector scatter photocoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Retina Centers, P.C., Northwest Location, Tucson, Arizona
  - Retina Associates, SW, Tucson, Arizona
  - Jules Stein Institute, Los Angeles, California
  - Orange County Retina Associates, Santa Ana, California
  - New England Retina Associates, Hamden, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - The University of Chicago, Chicago, Illinois
  - Macula-Retina-Vitreous Service, Indianapolis, Indiana
  - Vitreo-Retinal Consultants & Surgeons, P.A., Wichita, Kansas
  - Retina Associates, New Orleans, Louisiana
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Center, Hagerstown, Maryland
  - New England Eye Center, Boston, Massachusetts
  - Massachusetts Eye & Ear Infirmary, Boston, Massachusetts
  - Lahey Clinic, The Eye Institute, Peabody, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Eye Foundation of Kansas City, Kansas City, Missouri
  - Charlotte Eye, Ear, Nose and Throat Associates, P.A., Charlotte, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Retina Associates of Cleveland Inc., Lakewood, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Casey Eye Institute, Portland, Oregon
  - Wills Eye Institute Retina Research, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Retina Research Institute of Texas, LLC, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - VitreoRetinal Consultants, Houston, Texas
  - Valley Retina Associates, P.A., McAllen, Texas
  - University of Wisconsin, Madison, Wisconsin
  - The Eye Institute, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Wroblewski JJ, Wells JA 3rd, Adamis AP, Buggage RR, Cunningham ET Jr, Goldbaum M, Guyer DR, Katz B, Altaweel MM; Pegaptanib in Central Retinal Vein Occlusion Study Group. Pegaptanib sodium for macular edema secondary to central retinal vein occlusion. Arch Ophthalmol. 2009 Apr;127(4):374-80. doi: 10.1001/archophthalmol.2009.14. PMID 19365011
- See also: Sponsor's Website — http://www.eyetech.com